CLINICAL TRIAL: NCT04891302
Title: A Double Blind, Randomized, Placebo-controlled, Multi-center, Proof of Concept Phase 2 Study to Evaluate the Safety and Efficacy of Clevudine in Patients Diagnosed With Mild and Moderate COVID-19
Brief Title: The Proof of Concept Phase 2 Study to Evaluate the Safety and Efficacy of Clevudine in Patients With Mild and Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK-CLV-203
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Clevudine
MeSH Terms: conditions — COVID-19 | interventions — clevudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clevudine (Experimental): Clevudine 150 mg once a day for 10 days
  Interventions: Drug: Clevudine
- Placebo (Placebo Comparator): Matching Placebo once a day for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clevudine — Clevudine 150mg (5 capsules) once a day will be administered orally and can be taken regardless of food intake for 10 days
  Arms: Clevudine
Drug: Placebo — Matching Placebo (5 capsules) once a day will be administered orally and can be taken regardless of food intake for 10 days
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to assess the safety and efficacy of Clevudine 150 mg versus placebo once daily administration with standard of care therapy for 10 days in patients with mild and moderate COVID-19.

ELIGIBILITY:
Key Inclusion Criteria:

1. Over 19 years of age
2. COVID-19 confirmed by a real-time RT-PCR tests, and hospitalized
3. Patients who experienced first symptom related to COVID-19 within 7days prior to enrollment and confirmed 2 or more relative symptoms at the time of randomization.
4. Patients with peripheral capillary oxygen saturation(SpO2) greater than 94% at the time of screening, who do not need supplemental oxygen therapy.

Key Exclusion Criteria:

1. Patients who participated in other clinical trials related to COVID-19
2. Patients who were administered drugs directly to COVID-19 24hours prior to the start of the study.
3. Patients who need oxygen supply or breathing device (non-invasive mechanical ventilation(via mask)), mechanical ventilator requirement (via endotracheal tube or tracheostomy tube, ECMO requirement) at the time of screening or baseline
4. Patients whose AST or ALT has increased by more than 5 times the normal lab value.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
The amount of SARS-CoV-2 virus reduction on Day 11 compared to the the baseline. | Day 11

SECONDARY OUTCOMES:
The time consumed for clinical improvement. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day 29 (or EOT)
The rate of subjects tested as negative SARS-CoV-2 in consecutive two days of Real-Time RT-PCR tests. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day 29 (or EOT)
The amount of SARS-CoV-2 virus reduction on Day 4, Day 8, Day 15, Day 22 and Day 29 compared to the the baseline. | Day 4, Day 8, Day 15, Day 22 and Day29 (or EOT)
The rate of subjects indicated by the improvement of lung invasive. | Within Day 29 (or EOT)
The cycle threshold values change from baseline. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day29
The viral load change from baseline. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day29
The C-reactive protein change from baseline. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day29
The procalcitonine change from baseline. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day29
The rate of subjects who received new oxygen supplement at visit after baseline. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day 29 (or EOT)
The time of subjects discharged from the hospital. | Day 4, Day 8, Day 11, Day 15, Day 22 and Day 29 (or EOT)

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Chungnam National University Hospital, Daejeon
  - Ajou University Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Myongji Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Incheon Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Medical Center, Seoul